CLINICAL TRIAL: NCT03055533
Title: A Feasibility Study of Headsprout Reading Program in Children With Autism Spectrum Disorder and Reading Delay
Brief Title: Headsprout Reading Program in Children With Autism Spectrum Disorder and Reading Delay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0275-18-EP
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Behavioral; Social; Headsprout reading program
MeSH Terms: conditions — Autism Spectrum Disorder; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention with Headsprout reading program (Experimental): Participants randomized to this study arm will begin treatment with the Headsprout program right away. Reading assessments will occur at the beginning and end of 12 weeks of treatment. Participation may be in clinic or via telehealth.
  Interventions: Behavioral: Headsprout reading program
- Delayed intervention (No Intervention): Participants randomized to this study arm will have reading assessments at the beginning and end of the study, but they will not begin treatment with the Headsprout program until after their participation in the study ends (12 weeks). Participation may be in clinic or via telehealth.

INTERVENTIONS:
Behavioral: Headsprout reading program — Headsprout is a commercially available, computer-based program reading intervention that can be tailored to meet the individual needs of each child. Participants will have treatment sessions with a trained therapist lasting one to two hours, two to four days a week, for approximately twelve weeks.
  Arms: Immediate intervention with Headsprout reading program

SUMMARY:
Headsprout is a commercially available computer-based reading program that teaches children fundamental reading skills, including phonics, fluency, and comprehension. The Headsprout reading intervention has been shown to be effective with children with various levels of reading skills, but it has not been rigorously tested in children with autism spectrum disorder (ASD). The purpose of this study is to evaluate the effectiveness of Headsprout in a pilot sample of 18 children with ASD and reading delays to serve as a foundation for a larger, future randomized clinical trial (RCT).

Eighteen participants will be included in the study and randomly assigned to one of two groups; the first group will immediately receive treatment with the Headsprout reading program and the second treatment group will receive treatment after 12 weeks. Treatment sessions will occur for one to two hours, two to four days a week, for twelve weeks. The participants who do not receive treatment immediately will be asked to complete reading assessments periodically throughout their wait time. Participation may occur in clinic or via telehealth.

DETAILED DESCRIPTION:
A large number of children with autism spectrum disorder (ASD) experience reading delays, yet few empirically supported reading interventions exist for this population. Reading delay can interfere with academic progress, impede vocational opportunities, hinder self-expression, and limit capacity for independent living. Accessing empirically supported interventions for reading skills can be difficult, with parents of children with ASD facing long waiting lists at specialty clinics, reflecting the simple fact that demand is greater than the supply of trained providers. There is a pressing need for access to affordable interventions that do not depend on specialty clinics.

As a commercially available, computer-based program, Headsprout may be a good fit for children with ASD. Headsprout has shown effectiveness in children with reading delay uncomplicated by ASD, but has not been rigorously studied in children with ASD. This study will investigate the effects of the Headsprout reading program on improving reading skills of children with autism. Eighteen children will be recruited and the researchers will evaluate their current language use by: 1) asking their parents to rate their child's language, 2) completing an echoic skill assessment. Current reading skills will be determined by administering a reading assessment that evaluates their reading accuracy and fluency.

Participants will be randomly assigned to one of two groups; the first group will immediately receive treatment with the Headsprout reading program and the second treatment group will receive treatment after 12 weeks. Participation may be in clinic or via telehealth. During the intervention, children will meet with a trained therapist, several times per week for approximately twelve weeks. The therapist will instruct them to complete various reading activities on the computer. These reading activities may include tasks such as receptively identifying letter names and letter sounds presented on the computer or practicing saying sounds out loud and blending combinations of sounds together.

The participants who do not receive treatment immediately will be asked to complete reading assessments periodically throughout their wait time. At the end of 12 weeks these participants will be able to start the Headsprout reading program.

ELIGIBILITY:
Inclusion Criteria:

* Age 7.0 to 18.9
* Confirmed clinical diagnosis of autism spectrum disorder (ASD)
* Minimum score of 40 on the Early Echoic Skills Assessment (EESA), which assesses language skills
* Minimum score of 20 on the Expressive Vocabulary Test (EVT), which assesses language skills
* Display deficits in reading, testing at least one grade levels below current grade level on the Dynamic Indicators of Basic Early Literacy Skills (DIBELS)
* English is primary language

Exclusion Criteria:

* Currently receiving an individualized intervention for reading
* Significant problem behavior

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Change in Kaufman Test of Educational Achievement score (KTEA-3) | Baseline and Week 12
  The Kaufman Test of Educational Achievement (KTEA™-3) measures academic achievement and identifies learning disabilities for children in pre-kindergarten through grade 12. The KTEA™-3 evaluates reading, math, written language and oral language. For this study we will only use the reading portion of this assessment.

SECONDARY OUTCOMES:
Change in the Dynamic Indicators of Basic Early Literacy Skills (DIBELS) assessment score | Baseline and Week 12
  The Dynamic Indicators of Basic Early Literacy Skills (DIBELS) assessment will be used to measure acquisition of early literacy skills, such as letter sounds, and oral reading fluency. The assessment provides a score for the number of letters read correctly per minute, the number of letter sounds read correctly per minute, the number of nonsense words read correctly per minute, and the number of words read correctly per minute. DIBELS is designed for children in kindergarten through 6th grade.

CONTACTS AND LOCATIONS:
Overall Officials: Bethany A Hansen, PhD, BCBA-D, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No